CLINICAL TRIAL: NCT06338787
Title: Novel Iron-Based Supplement for Active Young Women With Sub-Optimal Iron
Brief Title: A Novel Iron-Based Supplement for Athletes Aged 14-17
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Mitacs (Industry); Natural Sciences and Engineering Research Council, Canada (Other)
Responsible Party: Principal Investigator, Jane Shearer, Professor, University of Calgary
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-0826.2
Record Dates: First submitted 2024-03-24; First posted 2024-04-01 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Iron Deficiencies
Keywords: iron; microbiota; exercise
MeSH Terms: conditions — Iron Deficiencies; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Iron/yeast complex (FeSC) (Experimental): Iron Supplement
  Interventions: Other: FeSC

INTERVENTIONS:
Other: FeSC — Iron/yeast complex

SUMMARY:
Female endurance athletes are susceptible to iron deficiency and this can impact their exercise performance. This study aims to assess the efficacy of a novel iron supplement in improving iron status, gut microbiome, and exercise performance in endurance-trained females.

DETAILED DESCRIPTION:
Current iron supplements on the market are commonly associated with side effects including gastrointestinal distress, nausea, vomiting, and constipation. As a solution, the investigators have developed a novel delivery system for iron supplementation that overcomes many of these limitations. The goal of this study is to assess the efficacy of a yeast-iron complex in improving iron status, gut microbiome, and exercise performance in endurance-trained adolescent females (aged 14-17) with sub-optimal iron status. Participants will consume 40mg of elemental iron every second day for 8 weeks. Before and after supplementation, participants will be assessed for exercise capacity (VO2max), iron status, and the current state of the gut microbiome. each week during supplementation, participants will complete a survey in which they will report feelings of stress and recovery as well as gastrointestinal symptoms.

ELIGIBILITY:
Inclusion Criteria:

* cis-gendered female 14-18 years old
* sub-optimal iron status (ferritin ≤45mcg/ L)
* At least 1 year past the age of menarche
* Engage in moderate to vigorous endurance activity for at least 3 hours a week

Exclusion Criteria:

* Supplemented with iron iron (>5mg/day), prebiotics, or probiotics in last 3 months
* antibiotic use in last 3 months
* - Energy availability >30 kcal/kg lean body mass

Ages: 14 Years to 17 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2024-06-17 (Actual); Primary Completion 2025-03-12 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Iron Status | Baseline, 4 weeks, 8 weeks
  Ferritin
Hemoglobin | Baseline, 4 weeks, 8 weeks
  Hemoglobin concentration
Lower Gut microbiome | Baseline, 4 weeks, 8 weeks
  Fecal sample

SECONDARY OUTCOMES:
Exercise Capacity | Baseline, 4 weeks, 8 weeks
  Oxygen Consumption (VO2max)

OTHER OUTCOMES:
Gastrointestinal Symptoms 1 | Weekly for 8 weeks
  Gastrointestinal Symptoms Questionnaire (Scale 0-4; lower scores indicate reduced severity of symptoms)
Gastrointestinal Symptoms 2 | Weekly for 8 weeks
  Patient-Reported Outcomes Measurement Information System (Scale 0-4; lower scores indicate reduced severity of symptoms)
Sleepiness | Weekly for 8 weeks
  Epworth Sleepiness scale (scale 0-3; increased score indicates increased sleepiness)
Stress and Recovery | Weekly for 8 weeks
  The Recovery-Stress Questionnaire (scale 1-6; higher scores indicate better outcomes)

CONTACTS AND LOCATIONS:
Overall Officials: Jane Shearer, PhD, Principal Investigator — University of Calgary
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No